CLINICAL TRIAL: NCT00332566
Title: Immunogenicity, Reactogenicity & Safety of a Booster Dose of GSK Biologicals' DTPw-HBV/Hib Kft Vaccine Vs GSK Biologicals' DTPw-HBV/Hib Vaccine, in Infants Who Received a 3-Dose Primary Vaccination Course With the Same Vaccines.
Brief Title: Assess Immunogenicity, Reactogenicity, Safety of a Booster of GSK Biologicals DTPw-HBV/Hib Kft Compared to DTPw-HBV/Hib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106602
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B; Whole Cell Pertussis; Tetanus; Haemophilus Influenzae Type b; Diphtheria
MeSH Terms: conditions — Hepatitis B; Tetanus; Haemophilus Infections; Diphtheria

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: DTPw-HBV/Hib Kft vaccine GSK323527A
- Group B (Active Comparator)
  Interventions: Biological: Tritanrix™-HepB/Hiberix™

INTERVENTIONS:
Biological: DTPw-HBV/Hib Kft vaccine GSK323527A — Intramuscular injection, 1 dose
  Arms: Group A
Biological: Tritanrix™-HepB/Hiberix™ — Intramuscular injection, 1 dose
  Arms: Group B

SUMMARY:
This booster study will assess the immunogenicity, reactogenicity and safety of a booster dose of GSK Biologicals' DTPw-HBV/Hib Kft. vaccine versus DTPw-HBV/Hib vaccine, in healthy children, 18 to 24 months of age, who received the same vaccine for primary vaccination. Prior to the booster dose, this study will also assess the persistence of antibodies to the vaccine antigen components administered in the primary vaccination course. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female toddler, 18 to 24 months of age at the time of booster vaccination, who completed the three-dose primary vaccination course in the 101223 study.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 30 days after administration of the booster vaccine dose, with the exception of oral polio vaccine (OPV).
* Previous booster vaccination against diphtheria, tetanus, pertussis, hepatitis B and Hib disease since the conclusion visit of the 101223 study.
* History of diphtheria, tetanus, pertussis, hepatitis B and Hib disease.
* Known exposure to diphtheria, tetanus, pertussis, hepatitis B and Hib disease since the conclusion visit of the 101223 study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products during the study period.
* Other conditions which in the opinion of the investigator may potentially interfere with interpretation of study outcomes.
* One of the following adverse events that constitute absolute contraindications to further administration of DTP vaccine, having occurred after previous administration of DTPw vaccine.

  * Known hypersensitivity to any component of the vaccine, or having shown signs of hypersensitivity after previous administration of diphtheria, tetanus, pertussis or HB vaccines.
  * Encephalopathy
  * Axillary temperature of >= 40 °C/ rectal temperature >= 40.5 °C within 48 hours of vaccination.
  * Collapse or shock-like state within 48 hours of vaccination.
  * Persistent, inconsolable crying lasting >= 3 hours occurring within 48 hours of vaccination.
  * Seizures with or without fever occurring within 3 days of vaccination.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2006-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Anti-polyribosyl-ribitol-phosphate (PRP) antibody concentration | One month after the booster dose
Anti-hepatitis B surface antigen (HBs) antibody concentration | One month after the booster dose
Anti-diphtheria antibody concentration | One month after the booster dose
Anti-tetanus antibody concentration | One month after the booster dose

SECONDARY OUTCOMES:
Anti-Bordetella pertussis (BPT) antibody concentration | One month after the booster dose
Anti-PRP antibody concentration | Prior to the booster dose
Anti-HBs antibody concentration | Prior to the booster dose
Anti-diphtheria antibody concentration | Prior to the booster dose
Anti-tetanus antibody concentration | Prior to the booster dose
Anti-BPT antibody concentration | Prior to the booster dose
Occurrence of solicited symptoms | During the 4-day follow-up period after the booster dose
Occurrence of unsolicited symptoms | During the 31-day follow-up period after the booster dose
Occurrence of serious adverse events | During the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Capital Federal, Buenos Aires, Argentina
- GSK Investigational Site, León, Nicaragua

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Espinoza F, Tregnaghi M, Gentile A, Abarca K, Casellas J, Collard A, Lefevre I, Jacquet JM. Primary and booster vaccination in Latin American children with a DTPw-HBV/Hib combination: a randomized controlled trial. BMC Infect Dis. 2010 Oct 15;10:297. doi: 10.1186/1471-2334-10-297. PMID 20950456
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 106602 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106602 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106602 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106602 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106602 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106602 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register